CLINICAL TRIAL: NCT04876443
Title: Impact of COVID-19 Outbreak on the Alcohol Consumption in Patients With Alcohol-related Liver Disease
Brief Title: Impact of COVID-19 Outbreak on the Alcohol Consumption in Patients With Alcohol-related Liver Disease (ICoLD)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 284173
Record Dates: First submitted 2021-05-05; First posted 2021-05-06 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Alcohol-related Liver Disease; Alcohol Dependence; Alcohol Withdrawal; Addiction, Alcohol
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Alcohol-related liver disease
  Interventions: Diagnostic Test: Study questionnaire

INTERVENTIONS:
Diagnostic Test: Study questionnaire — Study questionnaire related to drinking behaviour

SUMMARY:
The lockdown consequent to Coronavirus outbreak has had a differential impact on the drinking behaviour on the general population. The impact is unknown on the people with underlying chronic liver disease related to alcohol as some of them may have complex psychosocial background. The alcohol consumption in people with Alcohol-related Liver Disease (ArLD) is either due to alcohol dependence or related to their lifestyle. Alcohol dependence is a chronic relapsing remitting condition and this is associated with 60% mortality at 5 years in people who continue drinking.

Recovery from alcohol-use disorder (AUD) has been made more difficult during lock-down because peer support meetings such as Alcoholics Anonymous (AA) have no longer been taking place; a majority of the residential rehabilitation centres have closed or are no longer accepting admissions (PHE, 2020) and the single detoxification unit in London has been requisitioned as a COVID-19 step-down facility.

The aim of the study is to understand the influence of lockdown on the craving of alcohol and severity of alcohol dependence in patients with ArLD. The results from the study will enable us to identify the factors influencing the drinking behaviour during lockdown and a subsequent impact on episodes of decompensation and mortality.

DETAILED DESCRIPTION:
ICoLD, is a collaborative study between the King's College Hospital and SLaM. This is an observational self-report questionnaire study. The study population will comprise of people with alcohol-related chronic liver disease attending the Liver Outpatients and those admitted to the King's College Hospital. The study groups will be people who were abstinent of alcohol and people who have had history of alcohol consumption prior to lockdown.

The study will ascertain drinking behaviour prior to lock down and during lock down/COVID restrictions. The study uses the Severity of Alcohol Dependence Questionnaire (SADQ) to ascertain the severity of physiological dependence and the Obsessive compulsive Drinking Scale (OCDS) to characterise craving. The SADQ, OCDS and detailed Alcohol history is usually collected as a standard of care in patients with AUD.

The study will also investigate factors that could influence drinking behaviour during lockdown such as access to alcohol, affordability, pub closure/less socialising, boredom, time to reflect on health and psycho-social factors. Data on drinking behaviour, SADQ score and OCDS will be collected at any future lockdowns.

Patients with ArLD will be identified from the Liver outpatients or approached during their Hospital admission. Approximately, 700 patients with ArLD are followed in the Liver outpatients. 200 patients will be enrolled during the lockdown period, considering drop outs and a proportion of patients not willing to participate in the study. The study population will be followed up for a year after the final lockdown/COVID restrictions are lifted. No statisticians were involved in planning this study as it is a pilot study to generate hypotheses regarding the drivers of changes in drinking in this population during lockdown.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years.
* People with alcohol related Liver disease

Exclusion Criteria:

* Patient lacks capacity to consent to the study, e.g. due to hepatic encephalopathy, alcohol-related brain damage, or pre-existing learning disability
* Aged <18 years old
* Patients unable to understand English
* Patients being considered for liver transplant

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with alcohol-related chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-10-08 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Episodes of Hepatic decompensation | 24 months

SECONDARY OUTCOMES:
Mortality | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver Studies, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No